CLINICAL TRIAL: NCT01622595
Title: A Non-interventional Observational Study of Infectious Complications in Cancer Patients
Brief Title: UARK 2009-99 A Non-interventional Observational Study of Infectious Complications in Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator has left the institution.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 112265
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Aspergillosis; Candidemia; C. Difficile
Keywords: Aspergillosis; Candidemia; Candidiasis; C. Difficile; cytomegalovirus; respiratory syncytial virus (RSV); Influenza; CONS
MeSH Terms: conditions — Aspergillosis; Candidemia; Candidiasis; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OBSERVATIONAL STUDY OF INFECTIOUS COMPLICATIONS IN CANCER PATIENTS

DETAILED DESCRIPTION:
A NON-INTERVENTIONAL, OBSERVATIONAL STUDY OF INFECTIOUS COMPLICATIONS IN CANCER PATIENTS

ELIGIBILITY:
Inclusion Criteria:

* cancer patients with Infections

Exclusion Criteria:

* No Infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients with Infections
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To study the incidence, risk factors, clinical presentation, diagnosis and prognostic factors of infectious complications in cancer patients | 3 years
  To study the incidence, risk factors, clinical presentation, diagnosis and prognostic factors of infectious complications in cancer patients

SECONDARY OUTCOMES:
incidence | 3 years
  To determine the overall incidence of different infections, including bacterial, fungal and viral infections in cancer patients receiving chemotherapy and / or hematopoietic stem cell transplantation.
  * To describe the natural history of such infections in cancer patients.
  * To monitor the adherence of Myeloma institute for research and therapy(MIRT) health care workers to the MIRT standard operational procedures (SOPs)
  * To identify risk factors for the development of specific infections.
  * To validate surrogate markers as early diagnostic tools for various infections.

CONTACTS AND LOCATIONS:
Overall Officials: Senu Apewokin, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States